CLINICAL TRIAL: NCT01784107
Title: A Phase Ib/II Trial of Belotecan and Ifosfamide in Patients With Extensive Disease of Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Eun Kyung Cho, Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-GIRBA-2550
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; belotecan; Ifosfamide
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — belotecan; Ifosfamide

ARMS (1):
- Belotecan and Ifosfamide (Experimental)
  Interventions: Drug: Belotecan and Ifosfamide

INTERVENTIONS:
Drug: Belotecan and Ifosfamide

SUMMARY:
Phase 1 : To evaluate MTD(Maximal tolerated dose)and DLT(Dose limiting Toxicity) of Belotecan and Ifosfamide.

Phase 2 : To analyse efficacy and toxicity of Belotecan and Ifosfamide.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed extensive disease of Small cell lung cancer
* no prior chemotherapy or radiotherapy for lung
* measurable lesion for RECIST
* over 18 years
* ECOG 0~2
* expected life span more than 3 months

Exclusion Criteria:

* acute or active infection
* uncontrolled cerebral nerve symptoms or metastasis
* significant myocardial infarction or cardiac disease within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-07; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
MTD (maximal tolerated dose) | one year

SECONDARY OUTCOMES:
DLT(dose-limiting toxicity) | one year

OTHER OUTCOMES:
Response rate | one year
PFS(Progression-Free-Survival) | one year
Overall Survival | one year
Number of participants with adverse events | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea